CLINICAL TRIAL: NCT01059552
Title: Phase I Study of the HDAC Inhibitor Vorinostat With Chemotherapy and Radiation Therapy for Treatment of Locally Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Treatment of Locally Advanced Non-Small Cell Lung Cancer (NSCLC)
Acronym: NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FER-TH-031; NCI-2010-01913 (Registry Identifier: NCI Clinical Trials Reporting Office)
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Locally Advanced Non-small Cell Lung Cancer
Keywords: lung cancer; locally advanced lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- vorinostat (Experimental): Dose escalation of vorinostat, cisplatin, pemetrexed and radiation
  Interventions: Drug: vorinostat

INTERVENTIONS:
Drug: vorinostat — vorinostat once daily for 12 weeks of therapy
  Other Names: Zolinza

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose of the combination of vorinostat, cisplatin, pemetrexed, and radiation therapy in patients with unresectable stage IIIA/IIIB non-small cell lung cancer.

DETAILED DESCRIPTION:
This phase I trial will escalate doses of the histone deacetylase inhibitor (HDAC) vorinostat to a chemoradiation platform for cisplatin, pemetrexed and radiation to a dose of 70Gy in NSCLC patients with unresectable IIIA and dry IIIB disease. The endpoint will be to determine MTD of the combination.

ELIGIBILITY:
Inclusion Criteria:

* biopsy proven non-squamous NSCLC with unresectable stage IIIA or dry IIIB disease.
* FEV1 >/= 1 liter
* ECOG PS 0 or 1
* Able to swallow and absorb enterally
* Measurable disease per RECIST 1.1
* Adequate organ and marrow function including calculated creatinine clearance >/= 60 mL/min hepatic enzymes and alk phos </= 2.5 X ULN.

Exclusion Criteria:

* Chemotherapy or radiotherapy </= 4 weeks prior to registration (6 weeks for nitrosureas)
* Active bleeding
* Known brain mets
* Prior thoracic radiotherapy that would lead to overlap with current radiation field.
* More than 10% weight loss in 6 months.
* Pancoast tumors, supraclavicular or contralateral hilar lymph node involvement
* Known HIV positive
* Prior treatment with an HDAC inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-12-16 (Actual); Primary Completion 2015-07-22 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
To assess that safety and maximally tolerated dose of vorinostat in combination with chemoradiation for unresectable locally advanced NSCLC. | toxicity assessments will occur weekly

SECONDARY OUTCOMES:
To investigate progression free survival. | CT/PET scans will be done after 12 weeks of therapy and at 12 week intervals until documented progression
To evaluate response rates with this combination | CT/PET will be done following 12 weeks of therapy.
To assess if pre-treatment tumor expression of TS, ERCC1 and HDAC1, 2, 3 are associated with response rate. | Archival tissue will be tested and correlated to response rates.

CONTACTS AND LOCATIONS:
Overall Officials: Ranee Mehra, MD, Principal Investigator — Fox Chase Cancer Center
Locations (3):
- United States (3):
  - Moffitt Cancer Center, Tampa, Florida
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina